CLINICAL TRIAL: NCT06754813
Title: Association Between Uric Acid / High Density Lipoprotein Ratio and Monocyte / High Density Lipoprotein Ratio with Diabetic Complications
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat Allah Gamal Abdelnaser, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: HDL Uric UHR monocyte MHR DM
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- group 1: Diabetic patients without any macrovascular and microvascular Complications.
- group 2: Diabetic patients with macrovascular (stroke, coronary heart disease, Peripheral artery disease) and microvascular (DN and DR) complications
- group 3: Apparent healthy subjects as control group.

SUMMARY:
Type 2 diabetes mellitus (T2DM) poses a formidable global health challenge, with complications arising in both the microvascular and macrovascular domains as glycemic control worsens.the aim of the study to evaluate uric acid / high density lipoprotein cholesterol ratio and monocyte / high density lipoprotein ratio in studied groups. Association between Uric Acid / high density lipoprotein cholesterol ratio and monocyte / high density lipoprotein cholesterol ratio and diabetic Complications (macrovascular and microvascular).

DETAILED DESCRIPTION:
Hemoglobin A1c (HbA1c) continues to serve as the primary retrospective marker to assess glycemic management, but the inability to monitor daily blood glucose fluctuations remains a persistent concern

Uric acid is the final enzymatic product of purine nucleoside and free base degradation. Elevated levels of serum uric acid (SUA) are widely recognized as a risk factor for macrovascular and microvascular complications. Hyperuricemia is particularly common in patients with hyperlipidemia.

It has been established that SUA levels are proportional to triglyceride (TG), total cholesterol (TC), and low-density lipoprotein (LDL) levels. SUA promotes the oxidation of LDL, which is considered to be a key event in atherosclerotic plaque formation. The findings of several epidemiological studies have thus provided evidence to indicate a clear independent association between elevated SUA levels and an increased incidence of atherosclerotic disease or mortality Decreased serum levels of High-density lipoprotein cholesterol (HDL-c) are proposed to be related to worse metabolic status and reduced HDL-c is even a marker of metabolic syndrome.

A combination of these two metabolic parameters uric acid to HDL-c ratio (UHR) which is a more useful predictor of metabolic deterioration High-density lipoprotein- cholesterol acts by reducing proinflammatory responses triggered by monocytes, effectively restricting monocyte proliferation, activation and migration, and plays a role in the anti-oxidant mechanism. In contrast, reduced levels of HDL-c in the blood stream imply a worsening metabolic profile and are a component of the metabolic syndrome Uric acid can cause atherosclerosis and insulin resistance by reducing nitric oxide production, promoting vascular smooth muscle proliferation, and resulting in endothelial dysfunction. Additionally, low levels of HDL-c play a role in the development of metabolic syndrome and insulin resistance.

More recently, the uric acid-to-HDL-c ratio (UHR) has been identified as a marker that increases in inflammatory conditions . Monocytes and macrophages play crucial roles in damage to pancreatic islet cells, islet inflammation and impaired insulin signaling in T2DM. The monocyte/ HDL-c ratio (MHR) has been proposed as an indicator of ongoing low-grade metabolic inflammation and has been suggested studies to be used as a marker for cardiovascular disease and chronic kidney disease .

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* age more than 18 years old
* both sex

Exclusion Criteria:

* Individuals with malignancies, pregnant women, those using furosemide, thiazide, acetylsalicylic acid, losartan group drugs, cholesterol lowering drugs, patients with other autoimmune disorders, patients with chronic kidney disease and gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic patients who attending the Diabetes Clinic of Internal Medicine Department, Assiut University Hospital from January 2025 till January 2026.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
uric acid / high density lipoprotein cholesterol ratio | baseline
  Calculation of UHR was calculated by dividing serum uric acid value by HDL-c value
monocyte / high density lipoprotein ratio | baseline
  calculated by dividing of count of monocyte by HDL-c level

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S20-S42. doi: 10.2337/dc24-S002. PMID 38078589